CLINICAL TRIAL: NCT03928015
Title: A Single Centre Randomized Controlled Trial To Evaluate Dronabinol For Acute Pain Management In Adults With Traumatic Injury
Brief Title: Evaluation of Dronabinol For Acute Pain Following Traumatic Injury
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This trial did not enroll subjects. After initial approval we procured an appropriate placebo. Before IRB the amendment was approved, the COVID-19 pandemic placed a hold on all non-essential research activity at the enrolling hospital.
Sponsor: CommonSpirit Health (Other)
Responsible Party: Principal Investigator, Claire Swartwood, Pharmacy Residency Program Director, CommonSpirit Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1382279
Record Dates: First submitted 2019-04-09; First posted 2019-04-25 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Traumatic Injury; Pain, Acute
Keywords: marijuana; dronabinol; morphine milligram equivalents
MeSH Terms: conditions — Wounds and Injuries; Acute Pain; Marijuana Abuse | interventions — Dronabinol; Standard of Care

STUDY DESIGN:
Intervention Model Description: Open label, randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adjunctive dronabinol (Experimental): Dronabinol 5mg BID and adjusting within the range of 2.5mg - 10mg BID, as an adjunct to systemic analgesics
  Interventions: Drug: Adjunctive dronabinol
- Systemic analgesics (Active Comparator): Systemic analgesics only
  Interventions: Drug: Systemic analgesics

INTERVENTIONS:
Drug: Adjunctive dronabinol — 5mg BID and adjusting within the range of 2.5mg - 10mg BID, minimum of 48 hours, as an adjunct to systemic analgesics
  Other Names: Marinol
  Arms: Adjunctive dronabinol
Drug: Systemic analgesics — multimodal analgesia including opioid and non-opioid analgesics
  Other Names: standard of care
  Arms: Systemic analgesics

SUMMARY:
Single center, non-blinded, randomized controlled trial. Enrollment is based on ≥50 MME within 24 hours of admission, followed by a 24 hour screening/randomization window and a participation period extending through the acute hospitalization period.

A total of 122 adult patients admitted with a traumatic injury will be randomized 1:1 across 2 study arms: adjunctive dronabinol or systemic analgesics only. Patients randomized to the dronabinol arm should receive their first dose within 12 hours of randomization; patients will also receive PRN as needed systemic analgesics for pain. Except for the analgesia protocol, all other interventions will be equivalent for participants in both arms.

The clinical effects of analgesia treatment arm will be evaluated during the acute hospitalization (hospital admission through discharge or death). The primary efficacy endpoint will be assessed starting at 48 hours after randomization and carried through to discharge.

DETAILED DESCRIPTION:
Single center, non-blinded, randomized controlled trial. Enrollment is based on ≥50 MME within 24 hours of admission, followed by a 24 hour screening/randomization window and a participation period extending through the acute hospitalization period.

A total of 122 adult trauma patients will be randomized 1:1 across 2 study arms: adjunctive dronabinol or systemic analgesics only. Patients randomized to the dronabinol arm should receive their first dose within 12 hours of randomization, starting with 5mg BID and adjusting within the range of 2.5mg - 10mg BID. Patients randomized to dronabinol will also receive PRN as needed systemic analgesics for pain. Except for the analgesia protocol, all other interventions are performed in the context of everyday clinical practice, and thus will be equivalent for participants in both arms.

The clinical effects of analgesia treatment arm will be evaluated during the acute hospitalization (hospital admission through discharge or death). The primary efficacy endpoint will be assessed starting at 48 hours after randomization and carried through to discharge.

The primary trial objective is to evaluate the efficacy of adjunctive dronabinol versus no adjunctive dronabinol (systemic analgesics only) on reduction in opioids in adult patients with traumatic injury.

The secondary trial objectives include: evaluation of the efficacy of dronabinol versus no dronabinol (systemic analgesics only) for pain numeric rating scale (NRS) scores, hospital length of stay, complications, and adverse effects associated with analgesia.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years to 65 years old (inclusive)
2. Index admission for traumatic injury
3. High initial morphine equivalent use ≥ 50 mg in the first 24 hours from admission
4. Willing to divulge habitual marijuana usage (yes or no. Yes, habitual/chronic usage; no, recreational, former, or never usage)

Exclusion Criteria:

1. Patients on a pain management agreement
2. Patients who are nil per os (NPO) at the time of randomization or are expected to be NPO within the next 48 hours
3. Patients who have received or are expected to receive neuraxial/locoregional blocks for pain within the next 48 hours
4. Known allergy or previous hypersensitivity reaction to dronabinol or sesame oil
5. Patients prescribed dronabinol between arrival and prior to screening/randomization
6. Pregnancy or breast feeding
7. Incarceration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
Morphine equivalent use | Post-randomization (48 hours after randomization) - pre-randomization (24 hours prior to randomization)
  Change in morphine milligram equivalent (MME) use

SECONDARY OUTCOMES:
Pain scores | Post-randomization (48 hours after randomization) - pre-randomization (24 hours prior to randomization)
  Change in pain numeric rating scale (NRS) score, which is on a scale of 0-10. A value of 0 indications no pain and a value of 10 indicates highest level of pain
Incidence of complications | Acute hospitalization period
  Analgesic complications and other hospital complications
LOS | Acute hospitalization period
  Hospital LOS

CONTACTS AND LOCATIONS:
Overall Officials: Claire J Swartwood, PharmD, Principal Investigator — Centura Health - St. Anthony Hospital
Locations (1):
- St. Anthony Hospital, Lakewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Swartwood C, Salottolo K, Madayag R, Bar-Or D. Efficacy of Dronabinol for Acute Pain Management in Adults with Traumatic Injury: Study Protocol of A Randomized Controlled Trial. Brain Sci. 2020 Mar 12;10(3):161. doi: 10.3390/brainsci10030161. PMID 32178232